CLINICAL TRIAL: NCT02997163
Title: A PHASE I OPEN-LABEL PHARMACOKINETICS AND SAFETY STUDY OF TALAZOPARIB (MDV3800) IN PATIENTS WITH ADVANCED SOLID TUMORS AND NORMAL OR VARYING DEGREES OF RENAL IMPAIRMENT
Brief Title: An Open-Label Pharmacokinetics and Safety Study of Talazoparib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDV3800-01; C3441001 (Other: Alias Study Number); 2016-002536-33 (EudraCT Number)
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Results first posted 2020-02-20 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (control, normal renal function) (Experimental)
  Interventions: Drug: Talazoparib
- Group B (mild renal impairment) (Experimental)
  Interventions: Drug: Talazoparib
- Group C (moderate renal impairment) (Experimental)
  Interventions: Drug: Talazoparib
- Group D (severe renal impairment) (Experimental)
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — Daily oral doses of talazoparib 0.5 mg
  Other Names: MDV3800; BMN673

SUMMARY:
This trial will investigate the pharmacokinetics (PK) and safety of talazoparib in patients with advanced solid tumors and impaired renal function.

DETAILED DESCRIPTION:
At the End of the Study, patients with no clinically significant toxicities, no contraindications to continue treatment with talazoparib, and no disease progression (underlying cancer progression) may be eligible to continue talazoparib treatment in a separate open-label extension study after discussion with the Principal Investigator and obtaining Sponsor permission. Sponsor decision to allow the patient to continue dosing with talazoparib in an open-label extension study will be based on potential overall benefit-risk, patient acceptance and other relevant criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form (by the patient or a legally acceptable representative as per the local regulations) obtained prior to initiation of any study-specific procedure and treatment.
2. Female or male of at least 18 years of age.
3. Histologically or cytologically confirmed advanced solid tumor with no available standard approved treatment options in the opinion of the Investigator
4. Eastern Cooperative Oncology Group (ECOG) Performance status (PS) ≤ 2.
5. Expected life expectancy of ≥ 3 months.
6. Able to swallow the study drug (no contra indication to oral agents).
7. Renal function at screening and enrollment as defined by the Modification of Diet in Renal Disease (MDRD) equation.
8. Patient has had no clinically significant change in renal status within 3 months prior to screening, according to Investigator's review of clinical patient records.
9. Patient is not currently on hemodialysis and/or peritoneal dialysis for management of chronic kidney disease or acute failure/conditions.
10. Patient has no unstable renal function, defined as a change in estimated glomerular filtration rate (eGFR) (calculated with the MDRD equation) of > 25% for patients with mild and moderate renal impaired or as a change in eGFR > 30% for patients with severe renal impaired, from screening to enrollment.
11. Adequate other organ function at screening and enrollment.
12. Female patients of childbearing potential must have a negative serum pregnancy test at screening, and must agree to use a highly effective birth control method from the time of the first dose of study drug through 45 days after the last dose of study drug.
13. Male patients must agree to use a condom when having sex with a pregnant woman or with a non-pregnant female partner of childbearing potential, from 21 days before the first dose of study drug through 105 days after last dose of study drug.
14. Female patients must not be breastfeeding at screening nor during the study participation until 45 days after the last dose of study drug.
15. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Treatment within 14 days or five half lives prior to enrollment with any type of systemic anticancer-therapy or any investigational drug, whichever is longer.
2. Have not recovered (recovery is defined as CTCAE grade ≤ 1) from the acute toxicities of previous anticancer standard or investigational therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements.
3. Major surgery within 28 days prior to enrollment.
4. Serious accompanying cardiac disorder.
5. Active known or suspected brain metastasis or active leptomeningeal disease undergoing or requiring treatment.
6. Symptomatic or impending spinal cord compression or cauda equina syndrome.
7. Has undergone a liver transplant, kidney transplant or nephrectomy.
8. Prior allergic reaction or severe intolerance (meeting the criteria for a serious adverse event, a grade 3 or 4 AE, or permanent treatment discontinuation) to a poly ADP ribose polymerase (PARP) inhibitor.
9. Known myelodysplastic syndrome.
10. Seropositive for human immunodeficiency virus (HIV).
11. Any serious or unstable medical condition that interferes with ability to tolerate treatment or assessments associated with the protocol.
12. Gastrointestinal disorder affecting absorption.
13. Known or suspected hypersensitivity to any of the talazoparib capsule components.
14. Any condition or reason that interferes with ability to participate in the study, tolerate treatment or assessments associated with the protocol, causes undue risk, or complicates the interpretation of safety data, in the opinion of the Investigator or Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (6):
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Durairaj C, Chakrabarti J, Ferrario C, Hirte HW, Babu S, Piha-Paul SA, Plotka A, Hoffman J, Shi H, Wang DD. The Effect of Renal Impairment on the Pharmacokinetics and Safety of Talazoparib in Patients with Advanced Solid Tumors. Clin Pharmacokinet. 2021 Jul;60(7):921-930. doi: 10.1007/s40262-020-00983-y. Epub 2021 Mar 9. PMID 33686631
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=MDV3800-01

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Renal Function: Participants with normal renal function (estimated glomerular filtration rate [eGFR] greater than or equal to [>=] 90 milliliter per minute per 1.73 square meter [mL/min/1.73m^2]) received 0.5 milligrams (mg) (2 capsules of 0.25 mg) of talazoparib daily, orally for 22 days.
- Mild Renal Impairment: Participants with mild renal function (eGFR >= 60 and less than or equal to [<=] 89 mL/min/1.73m^2) received 0.5 mg (2 capsules of 0.25 mg) of talazoparib daily, orally for 22 days.
- Moderate Renal Impairment: Participants with moderate renal function (eGFR >= 30 and <=59 mL/min/1.73m^2) received 0.5 mg (2 capsules of 0.25 mg) of talazoparib daily, orally for 22 days.
- Severe Renal Impairment: Participants with severe renal function (eGFR >= 15 and <= 29 mL/min/1.73m^2) received 0.5 mg (2 capsules of 0.25 mg) of talazoparib daily, orally for 22 days.
Period: Overall Study
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Started | 9 | 9 | 8 | 8
Completed | 8 | 9 | 8 | 7
Not Completed | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis included all participants who received any amount of talazoparib.
Groups:
- Normal Renal Function: Participants with normal renal function (eGFR >= 90 mL/min/1.73m^2) received 0.5 mg (2 capsules of 0.25 mg) of talazoparib daily, orally for 22 days.
- Mild Renal Impairment: Participants with mild renal function (eGFR >= 60 and >=89 mL/min/1.73m^2) received 0.5 mg (2 capsules of 0.25 mg) of talazoparib daily, orally for 22 days.
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 9 | 9 | 8 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (6.99) | 65.4 (9.13) | 65.3 (6.45) | 72.8 (13.60) | 65.4 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 5 | 22
  Male | 4 | 3 | 2 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 9 | 7 | 8 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 7 | 8 | 7 | 7 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Multiple Dose: Area Under the Concentration Time Curve From 0 to 24 Hours (AUC0-24) of Talazoparib
Description: AUC0-24 of talazoparib was defined as the area under the concentration time curve from time 0 to 24 hours post-dose.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 22
Population: Pharmacokinetic (PK) analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
nanogram*hour per milliliter | 94.88 (27) | 106.5 (40) | 135.7 (45) | 249.8 (30)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 112.20, 90% CI 2-sided [80.06 to 157.26]
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 142.98, 90% CI 2-sided [103.03 to 198.42]
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 263.32, 90% CI 2-sided [187.88 to 369.06]

2. Primary Outcome: Multiple Dose: Maximum Observed Plasma Concentration (Cmax) of Talazoparib
Description: Cmax was defined as the maximum observed plasma concentration of talazoparib.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 22
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
nanogram per milliliter | 8.609 (35) | 9.568 (58) | 11.33 (45) | 16.30 (34)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 111.13, 90% CI 2-sided [74.40 to 166.01]
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 131.57, 90% CI 2-sided [89.12 to 194.25]
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 189.32, 90% CI 2-sided [126.74 to 282.80]

3. Primary Outcome: Multiple Dose: Area Under the Curve From Time 0 to 24 Hours for Unbound (AUC0-24u) Talazoparib
Description: AUC0-24u for unbound talazoparib was defined as the area under the concentration time curve from time 0 to 24 hours post-dose.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 22
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
nanogram*hour per milliliter | 28.33 (32) | 33.59 (31) | 39.47 (47) | 81.17 (36)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 118.58, 90% CI 2-sided [83.85 to 167.70]
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 139.34, 90% CI 2-sided [99.53 to 195.06]
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 286.61, 90% CI 2-sided [202.66 to 405.33]

4. Primary Outcome: Multiple Dose: Maximum Observed Plasma Concentration for Unbound (Cmaxu) Talazoparib
Description: Cmaxu was defined as the maximum observed plasma concentration for unbound talazoparib.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 22
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
nanogram per milliliter | 2.570 (42) | 3.019 (47) | 3.295 (48) | 5.296 (30)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 117.45, 90% CI 2-sided [79.74 to 172.99]
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 128.22, 90% CI 2-sided [88.05 to 186.72]
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Superiority; Percent Ratio of Geometric Means = 206.07, 90% CI 2-sided [139.91 to 303.51]

5. Secondary Outcome: Single Dose: Area Under the Concentration Time Curve From 0 to 24 Hours (AUC0-24) of Talazoparib
Description: AUC0-24 of talazoparib was defined as the area under the concentration time curve from time 0 to 24 hours post-dose.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 1
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 7 | 7
nanogram*hour per milliliter | 17.51 (59) | 23.60 (47) | 21.96 (40) | 29.98 (25)

6. Secondary Outcome: Single Dose: Maximum Observed Plasma Concentration (Cmax) of Talazoparib
Description: Cmax was defined as the maximum observed plasma concentration of talazoparib.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 1
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
nanogram per milliliter | 2.133 (56) | 2.422 (29) | 2.862 (75) | 2.624 (66)

7. Secondary Outcome: Single Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Talazoparib
Description: Tmax was defined as the time to reach maximum observed plasma concentration of talazoparib.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 1
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
hours | 1.515 [0.500 to 2.00] | 1.000 [0.970 to 2.12] | 0.9900 [0.480 to 2.00] | 1.830 [0.500 to 8.00]

8. Secondary Outcome: Single Dose: Fraction of Unbound Drug (Fu) in Plasma in Talazoparib
Description: Fraction of unbound drug (fu) was defined as the ratio of unbound drug concentration to the total drug concentration.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 6
ratio | 31.74 (22) | 33.71 (14) | 28.77 (7) | 33.91 (19)

9. Secondary Outcome: Single Dose: Area Under the Curve From Time 0 to 24 Hour for Unbound (AUC0-24u) Talazoparib
Description: AUC0-24u for unbound talazoparib was defined as the area under the concentration time curve from time 0 to 24 hours for unbound talazoparib.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 7 | 6
nanogram*hour per milliliter | 5.555 (81) | 7.956 (35) | 6.262 (39) | 10.95 (28)

10. Secondary Outcome: Single Dose: Maximum Observed Plasma Concentration for Unbound (Cmaxu) Talazoparib
Description: Cmaxu was defined as the maximum observed plasma concentration for unbound talazoparib.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 6
nanogram per milliliter | 0.6772 (67) | 0.8168 (62) | 0.8229 (70) | 1.031 (43)

11. Secondary Outcome: Multiple Dose: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Talazoparib
Description: Tmax was defined as the time to reach maximum observed plasma concentration of talazoparib.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 22
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
hours | 1.500 [0.970 to 4.00] | 2.000 [0.500 to 4.00] | 1.490 [0.470 to 4.02] | 3.880 [0.500 to 8.00]

12. Secondary Outcome: Multiple Dose: Plasma Trough Concentration (Ctrough) of Talazoparib
Description: Ctrough was defined as plasma trough (predose) concentration of talazoparib.
Time Frame: Predose on Day 22
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
nanogram per milliliter | 2.172 (34) | 2.680 (52) | 3.893 (45) | 7.917 (44)

13. Secondary Outcome: Multiple Dose: Apparent Oral Clearance (CL/F) of Talazoparib
Description: Drug clearance is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 22
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
liters per hour | 5.270 (27) | 4.698 (40) | 3.687 (45) | 2.000 (30)

14. Secondary Outcome: Multiple Dose: Accumulation Ratio (Rac) of AUC (0-24)
Description: Accumulation ratio for AUC0-24 was calculated as area under the curve from time zero to 24 hours on Day 22 divided by area under the curve from time zero to 24 hours on Day 1.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8 to 12, and 24 hours post-dose on Day 1 and Day 22
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 7 | 7
ratio | 5.418 (59) | 4.510 (42) | 6.239 (38) | 8.330 (36)

15. Secondary Outcome: Multiple Dose: Fraction of Unbound Drug (Fu) in Plasma in Talazoparib
Description: Fraction of unbound drug (fu) was defined as the ratio of unbound drug concentration to the total drug concentration.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8-12, and 24 hours post-dose on Day 22
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
ratio | 29.85 (24) | 31.54 (10) | 29.09 (9) | 32.49 (30)

16. Secondary Outcome: Multiple Dose: Unbound Apparent Oral Clearance (CLu/F) of Talazoparib
Description: Clearance of unbound drug is a measure of the rate at which unbound drug is metabolized or eliminated by normal biological processes.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8-12, and 24 hours post-dose on Day 22
Population: PK analysis population included all participants who had at least 1 reportable talazoparib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 7
liters per hour | 17.66 (32) | 14.89 (31) | 12.68 (47) | 6.614 (36)

17. Secondary Outcome: Single Dose: Amount of Talazoparib Excreted Unchanged in Urine From Time 0 to 24 Hours (Ae 0-24)
Description: Ae 0-24 is the amount of drug excreted unchanged in urine from time 0 to 24 hours postdose.
Time Frame: 0 to 24 hours on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 6
milligram | 0.05452 (51) | 0.05430 (38) | 0.02765 (59) | 0.01901 (78)

18. Secondary Outcome: Single Dose: Percentage of Dose of Talazoparib Excreted in Urine From Time 0 to 24 Hours (Ae 0-24%) at Day 1
Description: Ae0-24% was defined as the amount of drug excreted in urine from time 0 to 24 hours expressed as percentage of administered dose.
Time Frame: 0 to 24 hours on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 6 | 7 | 8 | 6
percentage of dose | 10.91 (51) | 10.85 (38) | 5.532 (59) | 3.795 (78)

19. Secondary Outcome: Multiple Dose: Amount of Talazoparib Excreted in Urine From Time 0 to 24 Hours (Ae 0-24%)
Description: Ae 0-24 is the amount of drug excreted unchanged in urine from time 0 to 24 hours postdose.
Time Frame: 0 to 24 hours on Day 22
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 7 | 7 | 7
milligram | 0.2584 (23) | 0.2321 (20) | 0.1637 (54) | 0.2005 (34)

20. Secondary Outcome: Multiple Dose: Percentage of Talazoparib Excreted in Urine From Time 0 to 24 Hours (Ae 0-24 %) of Talazoparib at Day 22
Description: Ae 0-24% was defined as the amount of drug excreted in urine from time 0 to 24 hours, expressed as percentage of administered dose.
Time Frame: 0 to 24 hours on Day 22
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 7 | 7 | 7
percentage of dose | 51.66 (23) | 46.40 (20) | 32.78 (54) | 40.07 (34)

21. Secondary Outcome: Multiple Dose: Renal Clearance (CLr) of Talazoparib at Day 22
Description: Renal clearance was calculated as cumulative amount of drug excreted in urine during the 24 hours dosing interval (Ae) divided by area under the plasma concentration time-curve from time zero to 24 hours postdose.
Time Frame: 0 to 24 hours on Day 22
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 7 | 7 | 5
liters per hour | 2.738 (37) | 2.180 (57) | 1.330 (97) | 0.7094 (35)

22. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. Treatment-emergent were events between first dose of investigational product and up to 30 days after the last dose of investigational product (up to 52 days) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Population: Safety analysis included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 9 | 9 | 8 | 8
Participants
  TEAEs | 7 | 8 | 8 | 7
  SAEs | 1 | 0 | 0 | 2

23. Secondary Outcome: Number of Participants With Abnormalities in Physical Examination
Description: Physical examination included examination of the general appearance, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. Findings were considered to be abnormal based on investigator's decision.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Population: Safety analysis included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 9 | 9 | 8 | 8
Participants | 0 | 0 | 0 | 0

24. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) of Participants
Time Frame: Baseline, Day 8, Day 15, Day 22, Safety follow up (Day 52)
Population: Safety analysis included all participants who received any amount of talazoparib. Here, "number analyzed" signifies participants evaluable for specific rows.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 9 | 9 | 8 | 8
millimeters of mercury (mmHg)
  Baseline | 115.4 (13.19) | 124.3 (11.55) | 123.8 (11.63) | 133.6 (17.25)
  Change at Day 8 | 9.0 (17.29) | -6.7 (18.28) | -2.5 (8.50) | -7.3 (11.29)
  Change at Day 15 | 1.9 (13.48) | -6.8 (7.03) | -5.6 (4.87) | -2.9 (18.05)
  Change at Day 22 | 7.3 (15.72) | -7.3 (12.66) | 0.1 (7.90) | 1.0 (12.02)
  Change at Day 52: number analyzed (Participants) | 1 | 1 | 3 | 5
  Change at Day 52 | -3.0 (NA) — Standard deviation was not estimable due to 1 participant with SBP. | -42.0 (NA) — Standard deviation was not estimable due to 1 participant with SBP. | 4.3 (9.02) | -10.8 (18.75)

25. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) of Participants
Time Frame: Baseline, Day 8, Day 15, Day 22, Safety follow up (Day 52)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 9 | 9 | 8 | 8
mmHg
  Baseline | 69.8 (7.69) | 78.3 (8.38) | 69.8 (5.65) | 74.8 (14.10)
  Change at Day 8 | 5.4 (4.48) | -4.6 (10.48) | 2.8 (8.15) | -3.4 (9.96)
  Change at Day 15 | -0.2 (6.02) | -5.9 (6.62) | 0.4 (8.86) | -1.1 (11.37)
  Change at Day 22 | 3.4 (10.50) | -4.6 (6.13) | 5.5 (11.95) | -4.0 (8.18)
  Change at Day 52: number analyzed (Participants) | 1 | 1 | 3 | 5
  Change at Day 52 | 4.0 (NA) — Standard deviation was not estimable due to 1 participant with DBP. | -18.0 (NA) — Standard deviation was not estimable due to 1 participant with DBP. | 1.0 (6.00) | -1.0 (20.98)

26. Secondary Outcome: Change From Baseline in Heart Rate of Participants
Description: Heart rate was measured in terms of beats per minute.
Time Frame: Baseline, Day 8, Day 15, Day 22, Safety follow up (Day 52)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 9 | 9 | 8 | 8
beats per minute
  Baseline | 85.2 (11.23) | 81.6 (21.86) | 80.1 (11.54) | 77.4 (23.34)
  Change at Day 8 | 3.3 (9.18) | -0.2 (8.74) | 2.1 (12.22) | -4.6 (23.40)
  Change at Day 15 | 3.7 (8.60) | -4.3 (10.56) | -1.8 (11.11) | -1.9 (16.07)
  Change at Day 22 | -1.7 (11.86) | -8.0 (5.85) | -0.9 (10.38) | -7.4 (20.56)
  Change at Day 52: number analyzed (Participants) | 1 | 1 | 3 | 5
  Change at Day 52 | -10.0 (NA) — Standard deviation was not estimable due to 1 participant with change in heart rate. | -15.0 (NA) — Standard deviation was not estimable due to 1 participant with change in heart rate. | 1.7 (2.52) | -0.8 (8.04)

27. Secondary Outcome: Change From Baseline in Respiratory Rate of Participants
Description: Respiratory rate was measured in terms of breaths per minute.
Time Frame: Baseline, Day 8, Day 15, Day 22, Safety follow up (Day 52)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 9 | 9 | 8 | 8
breaths per minute
  Baseline | 17.6 (0.88) | 18.4 (0.88) | 18.3 (1.67) | 17.8 (4.71)
  Change at Day 8 | 0.2 (0.67) | -0.3 (1.58) | 0.5 (2.07) | -0.8 (4.40)
  Change at Day 15 | 0.9 (1.05) | -0.8 (1.72) | 0.0 (2.14) | -1.0 (4.00)
  Change at Day 22 | 0.2 (0.67) | -1.1 (1.36) | 0.6 (2.45) | -1.0 (4.00)
  Change at Day 52: number analyzed (Participants) | 1 | 1 | 3 | 5
  Change at Day 52 | 0.0 (NA) — Standard deviation was not estimable due to 1 participant with change in respiratory rate. | 1.0 (NA) — Standard deviation was not estimable due to 1 participant with change in respiratory rate. | 1.3 (2.31) | -1.4 (6.31)

28. Secondary Outcome: Change From Baseline in Body Weight of Participants
Time Frame: Baseline, Day 8, Day 15, Day 22, Safety follow up (Day 52)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 9 | 9 | 8 | 8
kilograms
  Baseline | 68.60 (14.651) | 69.12 (14.914) | 85.84 (20.221) | 66.79 (13.277)
  Change at Day 8: number analyzed (Participants) | 9 | 9 | 8 | 7
  Change at Day 8 | 0.16 (1.030) | -0.62 (0.424) | -0.26 (0.912) | -0.26 (1.834)
  Change at Day 15 | -0.17 (1.707) | -0.38 (1.045) | 0.05 (1.590) | -0.23 (2.371)
  Change at Day 22 | -0.43 (2.366) | -0.78 (1.058) | 0.04 (1.722) | -0.75 (3.189)
  Change at Day 52: number analyzed (Participants) | 1 | 1 | 3 | 5
  Change at Day 52 | 4.90 (NA) — Standard deviation was not estimable due to 1 participant with change in weight. | 0.70 (NA) — Standard deviation was not estimable due to 1 participant with change in weight. | -0.67 (2.122) | 2.88 (14.597)

29. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG parameters included pulse rate (PR) interval, QRS duration, QT interval and corrected QT interval using Fridericia's formula (QTcF). Abnormality criteria: 1) PR interval: greater than equal to (>=) 25 percent (%) increase when baseline >= 300 msec; 2) QRS duration: >=50% increase when baseline >=140 msec; 3) QT interval: >= 500 msec: 4) QTCF interval: QTc interval using Fridericia's formula (QTcF interval) >= 500 msec when baseline >= 60. IFB stands for increase from baseline.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Population: Safety analysis included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 9 | 9 | 8 | 8
Participants | 2 | 1 | 5 | 3

30. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory parameters: erythrocytes, hematocrit, hemoglobin, white blood cells, absolute neutrophil count, lymphocytes, platelets ; albumin, alkaline phosphatase, alanine aminotransferase, aspartate transaminase , bilirubin, bicarbonate, blood urea nitrogen , calcium, chloride, creatinine, gamma -glutamyl transferase, glucose, lactate dehydrogenase, sodium, phosphate, potassium, total protein, uric acid, follicle-stimulating hormone; international normalized ratio / prothrombin time [activated] partial thromboplastin time; Urinalysis (pH, specific gravity, protein, glucose, ketones, bilirubin, blood, leukocyte esterase); Serum pregnancy test; Serology for Human Immunodeficiency Virus (HIV). Number of participants with laboratory test abnormalities as per National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE) version 4.03 were reported: Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Population: Safety analysis included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 9 | 9 | 8 | 9
Participants
  Grade 1 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

31. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: As per ECOG, participant's performance status was measured on 5 point scale: 0=fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature, e.g., light housework, office work. 2= ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair: 5: dead.
Time Frame: Baseline, Safety follow up (Day 52)
Population: Safety analysis included all participants who received any amount of talazoparib. Here, "Number Analyzed" signifies participants who were evaluable at specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 9 | 9 | 8 | 8
Participants
  Baseline: ECOG: 0 | 3 | 2 | 1 | 1
  Baseline: ECOG: 1 | 4 | 7 | 5 | 4
  Baseline: ECOG: 2 | 2 | 0 | 2 | 3
  Baseline: ECOG: 3 | 0 | 0 | 0 | 0
  Baseline: ECOG: 4 | 0 | 0 | 0 | 0
  Day 52: number analyzed (Participants) | 1 | 1 | 4 | 5
  Day 52: ECOG: 0 | 0 | 0 | 0 | 0
  Day 52: ECOG: 1 | 1 | 0 | 3 | 2
  Day 52: ECOG: 2 | 0 | 1 | 1 | 1
  Day 52: ECOG: 3 | 0 | 0 | 0 | 1
  Day 52: ECOG: 4 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/9 | 0/8 | 1/8
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9 | 0/8 | 2/8
Other Adverse Events (participants affected / at risk) | 7/9 | 8/9 | 8/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=9) | Mild Renal Impairment (N=9) | Moderate Renal Impairment (N=8) | Severe Renal Impairment (N=8)
CONDITION AGGRAVATED (General disorders) | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=9) | Mild Renal Impairment (N=9) | Moderate Renal Impairment (N=8) | Severe Renal Impairment (N=8)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 1 | 1 | 2
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 2 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 3 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 1 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 4 | 0 | 3 | 2
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0 | 1
CHILLS (General disorders) | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 2 | 4 | 1 | 1
GAIT DISTURBANCE (General disorders) | 0 | 1 | 0 | 0
INJECTION SITE BRUISING (General disorders) | 0 | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0 | 0
PERIPHERAL SWELLING (General disorders) | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 1 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
SUNBURN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 2
BLOOD ALBUMIN DECREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 1
BLOOD POTASSIUM INCREASED (Investigations) | 0 | 0 | 0 | 1
EASTERN COOPERATIVE ONCOLOGY GROUP PERFORMANCE STATUS WORSENED (Investigations) | 0 | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 2 | 0 | 1
DYSGEUSIA (Nervous system disorders) | 0 | 1 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0 | 0
DYSURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT02997163/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02997163/SAP_001.pdf